CLINICAL TRIAL: NCT03810053
Title: Utilizing Technology to Promote Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 228815
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-07

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile App/Online Module (Experimental): Subjects will watch a short video containing information about cancers and benefits of uptake cancer prevention and early detection measures. Information regarding gender, age, smoking status, BMI and positive cancer history in family will be captured. Subjects will be provided with a list of cancer prevention and early detection measures based on the responses provided.
  Interventions: Behavioral: Mobile App/Online Module

INTERVENTIONS:
Behavioral: Mobile App/Online Module — Short didactic explainer video that will provide information about cancers and benefits of uptake of cancer prevention and early detection measures.

SUMMARY:
The goal of the program is to develop an online module/a health application for cell phones which will share didactic information regarding cancer prevention and early detection measures. These module/application will be developed, and be tested among volunteers for feedback. In the future, these module/application will be disseminated widely to address cancer health disparity particularly in Arkansas.

DETAILED DESCRIPTION:
The application or the online module will play a short didactic explanation video that will provide information about cancers and benefits of uptake of cancer prevention and early detection measures. It is currently unknown which method will be used, the online module or the application for the purpose. The study participants will be subjected to only one method (once the method have been finalized and created). The video content will engulf information about cervical, breast, colorectal and lung cancer prevention and early detection. After the video, the application or the module will capture information on gender, age, smoking status, body mass index and positive cancer history in family. Watching the video and answering the questions will take approximately 5 minutes. The study participants will download the application on their personal cell phones and the data collected will be linked to identifying information in case they choose to receive the compensation and opt for the 6-month follow-up. Based on the responses provided, and the age and the gender, the participants will be provided with a list of cancer prevention and early detection measure(s). A subset of the study participants from ARResearch (only those who have agreed for the 6-month follow-up) will be asked if they are willing to be contacted by the study staff after 6 ±1 months (from the date of enrollment in the study) to enquire if they received/adopted the screening measures(s) that were suggested based on their age, gender and family history. They will be asked whether it is OK to call and/or e-mail them for more information to better describe barriers to obtaining cancer prevention and screening measures.

ELIGIBILITY:
Inclusion Criteria:

* Any ARResearch volunteer
* 18 years or older in age
* Have access to a personal cell phone and/or computer

Exclusion Criteria:

* Unable to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayumi Nakagawa, Ph.D, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile App/Online Module
Started | 290
Completed | 290
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mobile App/Online Module
Number analyzed (Participants) | 290
Age, Customized [Number; unit: participants]
  18-29 | 63
  30-39 | 84
  40-49 | 76
  >/=50 | 67
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 200
  Male | 87
  Neither | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 239
  More than one race | 12
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 290

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants to Learn New Information
Description: Percentage of participants that indicated they learned something new about cancer prevention measures.
Time Frame: up to 6 Months
Population: 290 participants ages 18 and over.
Measure: Number; unit: percentage of participants
Arm/Group | Mobile App/Online Module
Number analyzed (Participants) | 290
percentage of participants | 38.6

2. Primary Outcome: Percentage of Participants to Identify Needed Interventions
Description: Percentage of participants that identified interventions that they have not yet adopted from the use of the health application.
Time Frame: up to 6 months
Population: 290 participants 18 and over.
Measure: Number; unit: percentage of participants
Arm/Group | Mobile App/Online Module
Number analyzed (Participants) | 290
percentage of participants | 41.4

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Mobile App/Online Module
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03810053/Prot_SAP_000.pdf